CLINICAL TRIAL: NCT07053696
Title: Randomized Phase 1 Study of Safety, Pharmacokinetics, Segmental Lung Deposition, and Digital Validation of a Breath-Actuated EDDIS Inhalation Delivery System Using 99mTc-DTPA in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety, and Lung Deposition of 99mTc-DTPA Delivered Via the EDDIS System in Healthy Volunteers
Acronym: EDDIS-PK
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Changing regulatory requirements requiring changes in study design. Participants were not enrolled
Sponsor: Andrey Petrov (Other)
Collaborators: Ruslan Lytvin (Unknown)
Responsible Party: Sponsor-Investigator, Andrey Petrov, Principal Investigator, Petrov, Andrey
Organization: Petrov, Andrey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDDIS-PK-01
Record Dates: First submitted 2025-03-21; First posted 2025-07-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Inhalation Device; Lung Deposition; Aerosol; Pulmonary Drug Delivery; Radiolabeled Aerosol; Technetium Tc 99m DTPA; Scintigraphy

STUDY DESIGN:
Intervention Model Description: All participants will receive a single inhaled dose of radiolabeled aerosol (99mTc-DTPA) via the EDDIS system under controlled conditions.
Masking Description: No masking will be applied. Participants, investigators, and outcomes assessors will be aware of the intervention, as this is a non-therapeutic, Phase 1 imaging and device validation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Inhalation of 99mTc-DTPA via EDDIS System (Experimental): This arm includes all participants receiving a single inhaled dose of 99mTc-DTPA (radiolabeled aqueous solution in 0.9% NaCl, 2 ml total volume, 500-800 µCi), administered via the portable, breath-actuated EDDIS-IDDS (Enhanced Digital Dose Inhalation Delivery System).
  The procedure includes real-time digital recording of inspiratory parameters and post-inhalation planar scintigraphic imaging at 0, 15, and 30 minutes to assess pulmonary deposition.
  Pharmacokinetic samples (blood and urine) are collected for systemic exposure analysis. No control or comparator arm is included.
  Interventions: Drug: Technetium-99m Diethylenetriaminepentaacetic Acid; Device: EDDIS-IDDS (Enhanced Digital Dose Inhalation Delivery System)

INTERVENTIONS:
Drug: Technetium-99m Diethylenetriaminepentaacetic Acid — Technetium-99m Diethylenetriaminepentaacetic Acid A single inhaled dose of 99mTc-DTPA in 0.9% sodium chloride solution, total volume 2 ml, with radioactivity of 500-800 µCi. The solution is radiolabeled only in the aqueous phase to allow gamma scintigraphic imaging of pulmonary deposition. Delivered via breath-actuated EDDIS system. The formulation includes a non-labeled microdose of perfluorocarbon emulsion to simulate clinical aerodynamic behavior.
  Other Names: 99mTc-DTPA
Device: EDDIS-IDDS (Enhanced Digital Dose Inhalation Delivery System) — Portable, maintenance-free breath-actuated inhalation delivery system with integrated digital sensors. Records real-time data including inspiratory volume, flow rate, duration, and breath-hold time. Provides controlled aerosol delivery and secure transmission of inhalation parameters to the clinical monitoring platform.
  Other Names: EDDIS digital inhaler, breath-actuated inhalation device

SUMMARY:
Device:

EDDIS-IDDS (Enhanced Digital Dose Inhalation Delivery System) - a portable, breath-actuated, digitally monitored system for precision delivery of inhaled agents with automated recording of inspiratory volume, flow, duration, and breath-hold parameters.

Drug:

99mTc-DTPA (technetium-99m diethylenetriaminepentaacetic acid) - administered in aqueous solution (0.9% NaCl), radiolabeled for gamma scintigraphic imaging.

Total dose: 500-800 µCi in 2 ml solution.

Administration:

Single-dose inhalation under supervision in a clinical setting.

DETAILED DESCRIPTION:
This Phase 1, single-center, open-label clinical study is designed to evaluate the safety, pharmacokinetics, inhalation dynamics, segmental lung deposition, and digital monitoring capabilities of the breath-actuated EDDIS-IDDS (Enhanced Digital Dose Inhalation Delivery System) when used to deliver a radiolabeled aqueous formulation containing 99mTc-DTPA and a microdose of perfluorocarbon emulsion.

The investigational aerosol is administered via a digitally controlled inhalation system that automatically triggers delivery based on the patient's inspiratory effort. The system continuously records real-time parameters including tidal volume, inspiratory flow rate, inhalation duration, and breath-hold time. These data are securely transmitted and stored for analysis, enabling high-resolution correlation between inhalation patterns and lung deposition outcomes.

The radiolabel (99mTc-DTPA) is confined to the aqueous phase of the aerosol. The perfluorocarbon emulsion is included to simulate the aerodynamic behavior of complex liquid formulations and to evaluate their interaction with the lung architecture under controlled inhalation conditions. Radiolabeling is not applied to the perfluorocarbon phase, ensuring imaging specificity and avoiding nonspecific signal interference.

Imaging will be performed using planar gamma scintigraphy at 0, 15, and 30 minutes post-inhalation. Anterior and posterior projections will be acquired to allow quantitative segmental lung analysis. Measurements will include total deposition, central vs. peripheral distribution, and temporal sedimentation characteristics.

In parallel, blood samples will be collected at 1, 2, and 4 hours post-dose to determine systemic pharmacokinetics of the radiolabeled tracer. Urine samples collected at 4 hours will be used to calculate cumulative renal excretion. Adverse events, vital signs, and laboratory parameters will be monitored for 24 hours post-inhalation to assess tolerability and safety.

This study aims to establish a validated digital platform for inhaled delivery research and serve as a reference model for future studies involving targeted pulmonary therapeutics and diagnostic aerosols.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Healthy adults with no clinically significant medical history
* Normal spirometry (FEV1 ≥ 80% predicted)
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m²
* No prior exposure to radiopharmaceuticals in the past 12 months
* Able and willing to comply with study procedures and provide written informed consent
* Current or past use of tobacco products or electronic nicotine delivery systems (e.g., e-cigarettes) is not an exclusion criterion

Exclusion Criteria:

* History of asthma, COPD, or other chronic respiratory conditions
* History of lung surgery, pulmonary embolism, or interstitial lung disease
* Any ongoing respiratory infection or fever ≥ 38.0°C at screening or study day
* Uncontrolled or progressive arterial hypertension
* Known cardiovascular disease (e.g., arrhythmia, ischemic heart disease, heart failure)
* Presence of blood in saliva, hemoptysis, or any known pulmonary bleeding
* Diagnosed pulmonary emphysema
* Known coagulation disorders or use of anticoagulant therapy
* History of hypersensitivity to perfluorocarbons, DTPA, or radiopharmaceutical agents
* Prior exposure to radiopharmaceuticals within the last 12 months
* Participation in another clinical trial within the last 60 days
* Pregnancy or breastfeeding
* Use of any investigational or prescription drug within 30 days prior to study drug administration
* Any condition which, in the opinion of the investigator, would pose a health risk or interfere with study interpretation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Segmental lung deposition of 99mTc-DTPA measured by planar gamma scintigraphy | Within 30 minutes post-inhalation
  Quantitative analysis of 99mTc-DTPA distribution in lung segments using planar gamma scintigraphy imaging system with anterior/posterior views at 0, 15, and 30 minutes post-dose. Results expressed as percentage of total deposited dose per lung segment.
Incidence of treatment-emergent adverse events (TEAEs) assessed by clinical evaluation | Within 24 hours post-inhalation
  Number and severity of adverse events recorded after a single inhalation of 99mTc-DTPA via the EDDIS system, assessed through standardized clinical observation checklist, vital signs monitoring (blood pressure, heart rate, respiratory rate, temperature), and structured subject symptom reports using Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Radioactivity concentration in venous blood samples measured using gamma counter to determine systemic absorption of inhaled 99mTc-DTPA over time. Results expressed as counts per minute per milliliter (cpm/mL) | Up to 4 hours post-dose (samples at 1, 2, and 4 hours)
  Radioactivity in venous blood samples to determine systemic absorption of inhaled 99mTc-DTPA over time
Cumulative urinary excretion of 99mTc-DTPA measured by gamma counter analysis | up to 4 hours post-dose
  Total radioactivity in collected urine samples measured using gamma counter to estimate renal elimination of 99mTc-DTPA. Results expressed as percentage of administered dose excreted
Digital accuracy of inspiratory parameter recording assessed by calibration comparison | During inhalation procedure (real-time measurement)
  Comparison of EDDIS-recorded inspiratory volume (mL), flow rate (L/min), inhalation time (seconds), and breath-hold duration (seconds) with reference calibration measurements using validated spirometry equipment. Accuracy expressed as percentage deviation from reference values.

OTHER OUTCOMES:
Technical validation of the EDDIS inhalation delivery system performance assessment | During and immediately after inhalation (0-30 minutes)
  Technical validation checklist evaluating EDDIS breath-actuated system including real-time functionality assessment, data transmission integrity verification using signal processing analysis, and performance consistency evaluation across all subjects. Includes assessment of data completeness percentage, device startup response time (seconds), and fault/error detection system functionality using standardized device testing protocols.
Aerodynamic performance evaluation using particle size distribution analysis | During inhalation procedure (0-10 minutes)
  Evaluation of the impact of internal device architecture, aerosol path geometry, and mouthpiece design on aerosol dispersion using cascade impactor analysis, particle behavior assessment using laser diffraction particle size analyzer, and intrapulmonary airflow measurement using computational fluid dynamics modeling during breath-actuated delivery. Results expressed as mass median aerodynamic diameter (MMAD) and geometric standard deviation (GSD).
Inspiratory effort modulation and control assessment using digital sensor analysis | Real-time during inhalation procedure (0-10 minutes)
  Quantitative analysis using EDDIS digital sensor data to assess the system's ability to detect, monitor, and respond to variations in inspiratory intensity and breath profile in real time. Measurements include minimum activation threshold determination (L/min), dose delivery consistency evaluation under variable user effort (coefficient of variation), and real-time response accuracy assessment using pressure transducer validation

CONTACTS AND LOCATIONS:
Locations (1):
- Andrey Petrov Dr, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
This is a non-therapeutic, device validation study with radiolabeled imaging in healthy volunteers. No individual-level participant data will be shared. Aggregated, de-identified study results may be published in scientific journals or presented at scientific meetings.